CLINICAL TRIAL: NCT05074186
Title: Assessing the Safety and Effectiveness of a Neurological Thrombectomy Medical Device for Acute Ischemic Stroke
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Jacobs institute (Other)
Collaborators: University at Buffalo (Other)
Responsible Party: Principal Investigator, Adnan Siddiqui, Principal Investigator, Jacobs institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: DELPHI D001-PRT21-026
Record Dates: First submitted 2021-09-29; First posted 2021-10-12 (Actual); Last update posted 2025-09-15 (Actual); Status verified 2025-09

CONDITIONS: Ischemic Stroke
MeSH Terms: conditions — Ischemic Stroke

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (1):
- neurological thrombectomy device (Experimental): Revascularization device is an investigational device.
  Interventions: Device: neurological thrombectomy device is an investigational device.

INTERVENTIONS:
Device: neurological thrombectomy device is an investigational device. — Revascularization device is an investigational device.

SUMMARY:
The Jacobs Institute is participating in a Sponsor Investigator study designed to collect prospective clinical evidence to evaluate the use of a neurological thrombectomy device for clot retrieval in acute ischemic patients

DETAILED DESCRIPTION:
The neurological thrombectomy device is an investigational device

ELIGIBILITY:
Inclusion Criteria:

at least 18 years of age at time of consent Has baseline National Institutes of Health Stroke Scale (NIHSS) ≥ 8; Able to be treated within 8 hours of stroke symptom onset or Last Known Normal (LKN);

Exclusion Criteria:

Cannot provide consent or legally authorized representative not available to provide consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2021-06-08 (Actual); Primary Completion 2024-07-30 (Actual); Study Completion 2024-07-30 (Actual)

PRIMARY OUTCOMES:
Evaluate technical efficacy outcomes with radiographical measurements | Day 1
  The occurrence of all serious adverse device effects up to 90-days post-procedure Modified Thrombolysis in Cerebral Infarction (mTICI) score
outcomes with radiographical measurements | day 1
  The occurrence of all serious adverse device effects up to 90-days post-procedure Modified Thrombolysis in Cerebral Infarction (mTICI) score

SECONDARY OUTCOMES:
Evaluate technical efficacy outcomes with radiographical measurements | Day 3
  The occurrence of all serious adverse device effects up to 90-days post-procedure Modified Thrombolysis in Cerebral Infarction (mTICI) score
Evaluate technical efficacy outcomes with radiographical measurements | 90 days
  The occurrence of all serious adverse device effects up to 90-days post-procedure Modified Thrombolysis in Cerebral Infarction (mTICI) score

CONTACTS AND LOCATIONS:
Locations (1):
- kaledia Health/Buffalo General Medical Center/GVI, Buffalo, New York, United States

IPD SHARING:
Plan to Share IPD: No